CLINICAL TRIAL: NCT01523418
Title: Xarelto in the Prophylaxis of Post Surgical Venous Thromboembolism After Elective Major Orthopedic Surgery or Hip or Knee in Indian Patients
Brief Title: Study to Observe Safety of Xarelto in VTE Prophlylaxis After Elective TKR (Total Knee Replacement) or THR (Total Hip Replacement)
Acronym: XYRIS
Status: Withdrawn | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 15871; XA1111IN (Other: Company Internal)
Record Dates: First submitted 2012-01-30; First posted 2012-02-01 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Prophylaxis, Thromboembolism, Venous; Total Knee Replacement; Total Hip Replacement
Keywords: Xarelto; Thromboembolism, Venous; Orthopedic surgery; Factor Xa inhibitor; Observational study
MeSH Terms: conditions — Thromboembolism; Venous Thromboembolism | interventions — Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — The treatment with Xarelto 10mg tablets should comply with the recommendations. Rivaroxaban 10mg OD, 6-10 hours post-op, provided hemostasis has been achieved, for a period of 2 weeks (TKR) & 5 weeks (THR)

SUMMARY:
The primary objective of this study is to evaluate the safety of Xarelto in the prophylaxis of VTE in Indian patients undergoing elective TKR/THR

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of either sex, undergoing elective THR/TKR, in whom, Rivaroxaban is given for thromboprophylaxis
* Patients willing to give a written informed consent

Exclusion Criteria:

* Exclusion criteria must be read in conjunction with the local product information
* Patients on UFH / LMWH therapy, fondaparinux and vitamin K antagonists are not eligible.
* Patients with history of hypersensitivity to active ingredients or excipient :cellulose microcrystalline, croscarmellose sodium, lactose monohydrate, magnesium stearate, sodium lauryl sulfate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective TKR / THR
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Safety related variables are bleeding events reported as major or non-major adverse events | 3 months after the day of surgery
Symptomatic thromboembolic events (Deep vein thrombosis, Pulmonary embolism) reported as adverse events | 3 months after the day of surgery
All cause mortality | 3 months after the day of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer